CLINICAL TRIAL: NCT06478095
Title: Preoperative Visual Aids on Patients With Low Educational Backgrounds Undergoing Glaucoma Filtration Surgery
Brief Title: Preoperative Visual Aids on Glaucoma Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong (Other)
Collaborators: Shantou University Medical College (Other)
Responsible Party: Principal Investigator, Laiwen Lv, Mr., Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EC 20220505(4)-P30
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Anti-Glaucoma Medications
Keywords: Preoperative visit;glaucoma;filtering surgery
MeSH Terms: interventions — Audiovisual Aids

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: surgeons were blinded to the patient group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional oral education group (No Intervention): Patients were only orally educated about glaucoma, preoperative preparation, surgical procedures, anaesthesia methods, and precautions during the preoperative visit.
- The Visual aids plus conventional oral education group (Experimental): Patients were orally educated about glaucoma, preoperative preparation, surgical procedures, anaesthesia methods, and precautions with pictures and videos during the preoperative visit.
  Interventions: Behavioral: Visual aids

INTERVENTIONS:
Behavioral: Visual aids — Diagrams, models, and videos
  Arms: The Visual aids plus conventional oral education group

SUMMARY:
This study aims to evaluate the impact of preoperative visual aids on anxiety and pain management in patients with low educational backgrounds undergoing glaucoma filtration surgery.

DETAILED DESCRIPTION:
A randomized, single-blinded, single-centre clinical trial was conducted at a tertiary eye hospital in Shantou, China. Patients scheduled for glaucoma filtration surgery were randomly assigned to either a conventional oral education group or a visual aids group. Anxiety levels, pain scores, blood pressure, and pulse rates were measured at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients with age ≥18 years
* Illiterate or with ≤ 9 years of compulsory education
* Indications for filtering surgery

Exclusion Criteria:

* Mental illness
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Anxiety levels, pain scores, blood pressure, and pulse rates | 1 day prior to surgery; 30 minutes prior to surgery; 5 minutes after the onset of surgery; the conclusion of the surgical procedure
  measured at multiple time points

CONTACTS AND LOCATIONS:
Overall Officials: Chukai Huang, PhD, Study Director — Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong
Locations (1):
- Joint Shantou International Eye Center of Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data can be requested and accessed by contacting the study management teams of the studies on reasonable request. Such requests are adjudicated on a case-by-case basis. The study protocol and statistical analysis plan will be available and be accessed once the paper is accepted.